CLINICAL TRIAL: NCT00359268
Title: Identification of Novel Viruses
Brief Title: Identification of Viruses Associated With Diseases of Unknown Cause
Status: Terminated | Type: Observational
Why Stopped: Slow/insufficient accrual
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 010161; 01-I-0161
Record Dates: First submitted 2006-08-01; First posted 2006-08-02 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Viral Diseases
Keywords: Polymerase Chain Reaction; Random Priming; Nucleic Acid; Viral Genome
MeSH Terms: conditions — Virus Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: Any patient with a condition or disease whose etiology is unknown.

SUMMARY:
This study will try to identify new or known viruses responsible for diseases or conditions of unknown cause. Viruses are an important cause of illness. They have been identified as causes of several cancers, including certain liver cancers and cervical cancer. Several diseases, such as Kawasaki s disease, aplastic anemia, aphthous ulcers, and certain fevers of unknown origin in immune suppressed patients are thought possibly to be due to viruses, but their cause has not yet been determined. This study will use very sensitive molecular techniques to try to identify new or known viruses in patients with conditions of unknown causes. This study does not involve any treatment.

Any patient with a condition or disease whose cause is unknown may be eligible for this study. A referral from a local physician is required for patients who wish to enroll in this study.

Participants will have blood samples drawn up to four times during the study. The total amount of blood drawn in any 6-week period will not exceed 50 milliliters (about 3-1/2 tablespoons) for adults and 5 ml (about 1/2 tablespoon) per kilogram (2.2 pounds) for children. In addition, body fluids, such as joint or spinal fluid, or tissue samples, such as biopsy specimens, obtained previously for medical purposes, may be obtained for testing.

The patient s doctor will be informed of any positive findings from the samples. Identification of a virus does not necessarily mean that the virus is causing the patient s condition or disease. Additional tests from many patients with similar diseases or conditions are required before a virus can be definitively associated with a disease. Similarly, failure to find a virus does not necessarily mean that the patient is not infected with a virus that is causing the condition, as the tests used in this study are imperfect and will not detect certain forms of viruses that can cause disease.

DETAILED DESCRIPTION:
Viral infections are an important cause of morbidity and mortality in hospitalized patients. Viruses have also been identified as the probable cause of a number of malignancies including hepatocellular carcinoma and cervical carcinoma. The purpose of this study is to identify novel viruses (or known viruses) that are associated with diseases whose etiology is unknown. Blood samples, body fluids, or discarded tissues (e.g. previous biopsy or autopsy material) saliva swabs, nasopharyngeal swabs, skin biopsies, or mucosal biopsies will be obtained from patients with clinical syndromes or diseases whose etiology is unknown. Highly sensitive assays using the polymerase chain reaction will be performed to attempt to identify novel or known viruses that might be present in the blood, body fluids, or tissues. Knowledge gained from this study could provide important insights into the cause of diseases whose etiology is presently unknown.

ELIGIBILITY:
* INCLUSION CRITERIA:

Any patient with a condition or disease whose etiology is unknown.

Adequate venous access.

EXCLUSION CRITERIA:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a condition or disease whose etiology is unknown.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2001-05-08 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2020-03-23 (Actual)

PRIMARY OUTCOMES:
The purpose of this protocol is to obtain blood, body fluids, skin or mucosal biopsies, or discarded pathologic specimens from patients with diseases or syndromes of unknown etiology. | Ongoing
  Experimental studies will be performed on blood, body fluids, or discarded tissue specimens. Better understanding of the diseases of unknown etiology, improved diagnostic tests, and possible new treatments for diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey I Cohen, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Choo QL, Kuo G, Weiner AJ, Overby LR, Bradley DW, Houghton M. Isolation of a cDNA clone derived from a blood-borne non-A, non-B viral hepatitis genome. Science. 1989 Apr 21;244(4902):359-62. doi: 10.1126/science.2523562.
- [Background] Chang Y, Cesarman E, Pessin MS, Lee F, Culpepper J, Knowles DM, Moore PS. Identification of herpesvirus-like DNA sequences in AIDS-associated Kaposi's sarcoma. Science. 1994 Dec 16;266(5192):1865-9. doi: 10.1126/science.7997879.
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2001-I-0161.html